CLINICAL TRIAL: NCT04162847
Title: Harnessing Mobile Technology to Reduce Mental Health Disorders in College Populations
Acronym: iAIM EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Palo Alto University (Other); University of Michigan (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Denise Wilfley, Scott Rudolph University Professor of Psychiatry, Medicine, Pediatrics, and Psychological & Brain Sciences, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201901073; R01MH115128 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-11-14 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders; Depressive Disorder; Eating Disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mobile Coached Intervention (Experimental): This group will receive access to the mobile intervention for 6 months. They will be assigned to the primary program (i.e., anxiety, depression, or eating disorders) they screen positive for. If a person screens positive for more than one disorder, they will be given the choice of which program they want to start with. They will also be provided preventive interventions for anxiety, depressive, or eating of disorders they may not have but be at risk for. After two weeks in the program, the coach will assign the components presumed to be essential to intervention effects for comorbid disorder(s) and risk factors.
  Interventions: Device: SilverCloud Health Intervention
- Referral to Counseling Center (No Intervention): This group will receive information about how to make an appointment at their counseling center and will be encouraged to do so.

INTERVENTIONS:
Device: SilverCloud Health Intervention — SilverCloud Health is a mobile mental health platform offering cognitive-behavioral therapy-based guided self-help programs for preventing and treating anxiety, depression, and eating disorders as appropriate Participants in this arm will receive the support of a coach to guide them through the program. Participants will be able to communicate with their coach within the program.
  Arms: Mobile Coached Intervention

SUMMARY:
The prevalence of mental health problems among college populations has risen steadily in recent decades, with one third of today's students struggling with anxiety, depression, or an eating disorder (ED). Yet, only 20-40% of college students with mental disorders receive treatment. Inadequacies in mental health care delivery result in prolonged illness, disease progression, poorer prognosis, and greater likelihood of relapse, highlighting the need for a new approach for detecting mental health problems and engaging college students in services. The investigators have developed a transdiagnostic, low-cost mobile health targeted prevention and intervention platform that uses population-level screening for engaging college students in tailored services that address common mental health problems. This care delivery system represents an ideal model given its use of evidence-based mobile programs, a transdiagnostic approach that addresses comorbid mental health issues, and personalized screening and intervention to increase service uptake, enhance engagement, and improve outcomes. Further, this service delivery model harnesses the expertise of an interdisciplinary team of behavioral scientists, college student mental health scholars, technology researchers, and health economists. This work bridges the study team's collective leadership over the past 25 years in successfully implementing a population-based screening program in more than 160 colleges and demonstrating the effectiveness of Internet-based programs for targeted prevention and intervention for anxiety, depression, and EDs. Through this study, Investigators will test the impact of this mobile mental health platform for service delivery in a large-scale trial across a diverse range of U.S. colleges. Students who screen positive or at high-risk for clinical anxiety, depression, or EDs (excluding anorexia nervosa, for which more intensive medical monitoring is warranted) and who are not currently engaged in mental health services will be randomly assigned to: 1) intervention via the mobile mental health platform; or 2) referral to usual care (i.e., campus health or counseling center).

Participants in the study will be enrolled for 2 years and asked to complete surveys at baseline, 6 weeks, 6 months, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at participating colleges and universities who are 18 years old and older.
* Students who screen has high risk or clinical/subclinical for anxiety, depression, and, eating disorders.
* Students who are not currently in treatment, i.e., in the past month

Exclusion Criteria:

* Students who do not own a smartphone
* Students who are currently engaged in mental health treatment
* Students with anorexia nervosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6205 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilfley, PhD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Palo Alto University, Palo Alto, California
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Pennsylvania State University, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on the National Institute of Mental Health Data Archive as required by the National Institute of Health.
Time Frame: The data will be available at the end of the study, five years from now.
Access Criteria: The de-identified data will be shared on the National Institute of Mental Health Data Archive and will only be available to other researchers who have access to this platform.

REFERENCES:
- [Derived] Basterfield C, Fitzsimmons-Craft EE, Taylor CB, Eisenberg D, Wilfley DE, Newman MG. Internalizing psychopathology and its links to suicidal ideation, dysfunctional attitudes, and help-seeking readiness in a national sample of college students. J Affect Disord. 2024 Apr 1;350:255-263. doi: 10.1016/j.jad.2024.01.058. Epub 2024 Jan 13. PMID 38224742
- [Derived] Grammer AC, Vazquez MM, Fitzsimmons-Craft EE, Fowler LA, Rackoff GN, Schvey NA, Lipson SK, Newman MG, Eisenberg D, Taylor CB, Wilfley DE. Characterizing eating disorder diagnosis and related outcomes by sexual orientation and gender identity in a national sample of college students. Eat Behav. 2021 Aug;42:101528. doi: 10.1016/j.eatbeh.2021.101528. Epub 2021 May 15. PMID 34049053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
Started | 3103 | 3102
Completed 6-week Follow-up Assessment | 1386 | 1792
Completed 6-month Follow-up Assessment | 1363 | 1669
Completed 2-year Follow-up Assessment | 1627 | 1765
Completed | 3096 | 3101
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center | Total
Number analyzed (Participants) | 3103 | 3102 | 6205
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (4.0) | 20.2 (4.0) | 20.2 (4.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 802 | 811 | 1613
  Female | 2191 | 2179 | 4370
  Other | 110 | 112 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 519 | 527 | 1046
  Not Hispanic or Latino | 2584 | 2575 | 5159
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 35 | 42 | 77
  Asian | 473 | 466 | 939
  Native Hawaiian or Other Pacific Islander | 11 | 10 | 21
  Black or African American | 231 | 234 | 465
  White | 2134 | 2144 | 4278
  More than one race | 219 | 206 | 425
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3103 | 3102 | 6205
Diagnosis [Count of Participants; unit: Participants] — We assessed mental health diagnosis with brief validated measures.
  GAD-Q-IV for general anxiety. High risk score greater or equal to 5.7. Clinical: diagnostic criteria
  SPDQ for social anxiety. High risk score of 7.4+. Clinical: diagnostic criteria
  PDSR for panic disorder. High risk score of 8.8. Clinical: diagnostic criteria
  PHQ-9 for depression. High risk score of 5-9. Clinical score 10+
  SWED and WCS for eating disorders based on the last 3 months. High risk: weight concern score of 47+ and at least 1 purging episode. Clinical: 6 or more episode of binge eating or purging
  Participants
    High risk 0 clinical diagnosis | 839 | 828 | 1667
    1 clinical diagnosis | 752 | 824 | 1576
    2 clinical diagnosis | 710 | 656 | 1366
    3 clinical diagnosis | 538 | 540 | 1078
    4 clinical diagnosis | 231 | 218 | 449
    5 clinical diagnosis | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of the Mobile Mental Health Platform, Compared to Usual Care, in Changing the Number of Individuals With Mental Health Disorders.
Description: Effectiveness of the mobile mental health platform, compared to usual care, in reducing or preventing the number of individuals with mental health disorders (i.e., a positive screen for at least one of anxiety, depression, or eating disorder as the outcome reflecting a "clinical case"), assessed at 6 months and 2 years, with a primary endpoint of 2 years. Clinical case status will be determined using the Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) for generalized anxiety disorder, Social Phobia Diagnostic Questionnaire (SPDQ) for social anxiety disorder, the Panic Disorder Self Report (PDSR) for panic disorder, the Patient Health Questionnaire-9 (PHQ-9) for depression, and the Stanford-Washington University Eating Disorders Screen for eating disorders
Time Frame: baseline, 6 weeks, 6 months, and 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
Number analyzed (Participants) | 3103 | 3102
Participants
  Baseline: Number of participants with at least one clinical mental disorder | 2264 | 2274
  Baseline: Number of participants without any clinical mental disorder | 839 | 828
  6 weeks: Number of participants with at least one clinical mental disorder | 1764 | 1896
  6 weeks: Number of participants without any clinical mental disorder | 1339 | 1206
  6 month: Number of participants with at least one clinical mental disorder | 1743 | 1894
  6 month: Number of participants without any clinical mental disorder | 1360 | 1208
  2 year: Number of participants with at least one clinical mental disorder | 1723 | 1841
  2 year: Number of participants without any clinical mental disorder | 1380 | 1261
Statistical Analysis 1: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; Baseline; Test type: Superiority; p = .76, Regression, Logistic; Odds Ratio (OR) = .98, 95% CI 2-sided [.88 to 1.10]
Statistical Analysis 2: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; 6 week follow-up; Test type: Superiority; p = .001, Regression, Logistic; Odds Ratio (OR) = .84, 95% CI 2-sided [.76 to .93]
Statistical Analysis 3: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; 6 month follow-up; Test type: Superiority; p = .000, Regression, Logistic; Odds Ratio (OR) = .82, 95% CI 2-sided [.74 to .90]
Statistical Analysis 4: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; 2 year; Test type: Superiority; p = .002, Regression, Logistic; Odds Ratio (OR) = .86, 95% CI 2-sided [.77 to .95]

2. Secondary Outcome: Number of Participants Who Receive Treatment on the Mobile Mental Health Platform Compared to Number of Participants Who Receive Treatment in the Control Group.
Description: Uptake will be assessed as engaging in at least one session of mental health service use either online or in-person. This will be assessed based on actual use of the mobile program in the intervention condition and self-report of mental health services utilized or by reporting taking a new antidepressant or anti-anxiety medication in the control condition.
Time Frame: 6 weeks, 6 months, and 2 years
Population: Intervention: proportion of individuals who accessed the digital intervention platform during the 6 months post baseline period (this outcome was not relevant at 2 years for this condition).
  Control: proportion of individuals who, for 6 month and 2 year follow-up assessments, reported having had at least 1 session of counseling or psychotherapy or having started a new antidepressant or anti-anxiety medication (i.e., were not taking these medications at baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
Number analyzed (Participants) | 3103 | 3102
Participants
  6 month follow-up | 2308 | 938
  2 year follow-up: number analyzed (Participants) | 0 | 3102
  2 year follow-up |  | 1904
Statistical Analysis 1: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; A comparison of service uptake between the intervention and control groups over the 6-month follow-up period; Test type: Superiority; p = .000, Chi-squared; Odds Ratio (OR) = 6.70, 95% CI 2-sided [5.98 to 7.50]
Statistical Analysis 2: Comparison: Referral to Counseling Center; A secondary analysis using the same criterion for the intervention group (access to the digital intervention during the 6-month follow-up) but expanding the control group definition to include individuals who reported having psychotherapy or starting a new medication at any point during the full 2-year follow-up period; Test type: Superiority; p = .000, Chi-squared; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.64 to 2.04]

3. Secondary Outcome: Effectiveness of the Mobile Mental Health Platform, Compared to Usual Care, in Changing Disorder-specific Symptoms.
Description: Analyses will be conducted within each disorder subgroup separately. We will use the Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) for generalized anxiety disorder, this scale has a minimum value of 0 and a maximum value of 13, a lower score means a better outcome. The Social Phobia Diagnostic Questionnaire (SPDQ) for social anxiety disorder, this scale has a minimum value of 0 and a maximum value of 31, a lower score means a better outcome. The Panic Disorder Self Report (PDSR) for panic disorder, this scale has a minimum value of 0 and a maximum value of 24, a lower score means a better outcome. The Patient Health Questionnaire-9 (PHQ-9) for depression, this scale has a minimum value of 0 and a maximum value of 27, a lower score means a better outcome. The Eating Disorder Examination-Questionnaire (EDE-Q) for eating disorders, this scale has a minimum value of 0 and a maximum value of 6, a lower score means a better outcome.
Time Frame: baseline, 6 weeks, 6 months, and 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
Number analyzed (Participants) | 3103 | 3102
score on a scale
  PHQ-9 Baseline | 11.65 (5.91) | 11.68 (5.89)
  PHQ-9 6-week | 8.32 (5.52) | 9.43 (5.76)
  PHQ-9 6-month | 8.61 (5.95) | 9.29 (6.13)
  PHQ-9 2-year | 8.29 (5.79) | 8.73 (5.74)
  GADQ-IV Baseline | 6.56 (3.98) | 6.60 (3.94)
  GADQ-IV 6-week | 5.34 (3.84) | 5.73 (3.92)
  GADQ-IV 6-month | 5.43 (4.02) | 5.50 (4.02)
  GADQ-IV 2-year | 5.37 (3.96) | 5.49 (3.93)
  SPDQ Baseline | 12.44 (6.05) | 12.38 (6.06)
  SPDQ 6-week | 11.63 (6.16) | 12.06 (6.33)
  SPDQ 6-month | 11.20 (6.40) | 11.53 (6.41)
  SPDQ 2-year | 11.17 (6.30) | 11.40 (6.03)
  PDSR Baseline | 4.66 (6.96) | 4.72 (6.96)
  PDSR 6-week | 2.69 (5.75) | 2.84 (5.80)
  PDSR 6-month | 3.60 (6.41) | 3.62 (6.44)
  PDSR 2-year | 3.75 (6.60) | 3.82 (6.58)
  EDE-Q-Global Baseline | 1.81 (1.40) | 1.83 (1.39)
  EDE-Q-Global 6-week | 1.55 (1.24) | 1.74 (1.34)
  EDE-Q-Global 6-month | 1.48 (1.22) | 1.69 (1.33)
  EDE-Q-Global 2-year | 1.62 (1.29) | 1.67 (1.29)
Statistical Analysis 1: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PHQ-9 6 week; Test type: Superiority; p = .000, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 2: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PHQ-9 6 months; Test type: Superiority; p = .000, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 3: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PHQ-9 2 year; Test type: Superiority; p = .02, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 4: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; GADQ-IV 6 week; Test type: Superiority; p = .002, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 5: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; GADQ-IV 6 month; Test type: Superiority; p = .80, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 6: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; GADQ-IV 2 year; Test type: Superiority; p = .51, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 7: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; SPDQ 6 week; Test type: Superiority; p = .004, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 8: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; SPDQ 6 month; Test type: Superiority; p = .02, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 9: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; SPDQ 2 year; Test type: Superiority; p = .09, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 10: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PDSR 6 week; Test type: Superiority; p = .66, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 11: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PDSR 6 month; Test type: Superiority; p = .85, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 12: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; PDSR 2 year; Test type: Superiority; p = .97, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 13: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; EDE-Q Global 6 week; Test type: Superiority; p = .000, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 14: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; EDE-Q Global 6 month; Test type: Superiority; p = .000, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 15: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; EDE-Q Global 2 year; Test type: Superiority; p = .54, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions

4. Secondary Outcome: Effectiveness of the Mobile Mental Health Platform, Compared to Usual Care, in Changing Quality of Life and Functioning.
Description: Impairment/quality of life will be assessed using the Short Form-12 Health Survey. This scale has a minimum value of 0 and a maximum value of 100, a higher score means a better outcome for both the physical component and mental component.
Time Frame: baseline, 6 months, and 2 years
Population: Analysis we ran separately for the mental component summary (MCS) and the physical component summary (PCS).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
Number analyzed (Participants) | 3103 | 3102
score on a scale
  MCS Baseline | 34.11 (10.73) | 33.89 (10.69)
  MCS 6 months | 36.41 (11.49) | 35.95 (11.63)
  MCS 2 years | 37.85 (11.33) | 36.93 (11.40)
  PCS Baseline | 53.65 (7.63) | 53.85 (7.30)
  PCS 6 months | 63.21 (8.55) | 53.43 (8.31)
  PCS 2 years | 53.15 (7.84) | 53.42 (7.87)
Statistical Analysis 1: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; Mental component summary 6 months; Test type: Superiority; p = .48, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 2: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; Mental component summary 2 years; Test type: Superiority; p = .04, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 3: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; Physical component summary 6 months; Test type: Superiority; p = .97, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions
Statistical Analysis 4: Comparison: Mobile Coached Intervention vs Referral to Counseling Center; Physical component summary 2 years; Test type: Superiority; p = .80, multilevel modeling methods; Multilevel modeling was used to examine differences in changes in each outcome measure between the two conditions

5. Other Pre Specified Outcome: Examine if the Mobile Intervention Changes Avoidance for Individuals With or at High Risk for Anxiety and if Changes in Avoidance Are Associated With Clinical Benefit.
Description: Avoidance will be measured using item 3 of the Overall Anxiety and Impairment Scale.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Examine if the Mobile Intervention Changes Behavioral Activation for Individuals With or at High Risk for Depression and if Changes in Behavioral Activation Are Associated With Clinical Benefit.
Description: Behavioral activation will be measured using the Behavioral Activation for Depression Scale Short-Form.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Examine if the Mobile Intervention Changes Dietary Restraint and Weight/Shape Concerns for Individuals With or at High Risk for Eating Disorders and if Changes in Dietary Restraint and Weight/Shape Concerns Are Associated With Clinical Benefit
Description: Dietary restraint will be measured using the Eating Disorder Examination-Questionnaire Restraint subscale and change in weight/shape concerns using the Weight Concerns Scale.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Examine if the Mobile Intervention Changes in Dysfunctional Cognitions and if Changes in Dysfunctional Cognitions Are Associated With Clinical Benefit.
Description: Change in dysfunctional cognition will be measured using the Dysfunctional Attitude Scale Short form-2.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Examine if the Mobile Intervention Changes Cognitive-behavioral Therapy (CBT) Skills and if Changes in CBT Skills Are Associated With Clinical Benefit.
Description: Change in CBT skills will be measured using the self-report version of the Skills of Cognitive Therapy Scale.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Identify Other Putative Mediators of Change.
Description: To identify other putative mediators of change we will look at early engagement in help services, number of sessions completed, and rapid response.
Time Frame: baseline, 6 weeks, 6 months, 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months following the baseline.
Arm/Group | Mobile Coached Intervention | Referral to Counseling Center
All-Cause Mortality (participants affected / at risk) | 0/3103 | 0/3102
Serious Adverse Events (participants affected / at risk) | 0/3103 | 0/3102
Other Adverse Events (participants affected / at risk) | 0/3103 | 0/3102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT04162847/Prot_SAP_001.pdf